CLINICAL TRIAL: NCT00803608
Title: Prospective, Randomized, Multiple Site Clinical Trial Comparing the Effectiveness of Novel Pressure Based Insoles to Current Care For Ulcer Prevention
Brief Title: The CareFUL Prevention Trial
Acronym: CareFULPrevent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DIApedia, LLC (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DK05907405A1; R44DK059074 (NIH)
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Plantar Ulcer; Diabetes; Neuropathy Causing Loss of Protective Sensation
Keywords: Plantar; Ulcer; Diabetes
MeSH Terms: conditions — Foot Ulcer; Diabetes Mellitus; Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 02 (Active Comparator): Current standard of care insole
  Interventions: Device: Current standard of care insole
- 01 (Experimental): TrueContour® insole
  Interventions: Device: TrueContour® Insole

INTERVENTIONS:
Device: TrueContour® Insole — Novel designed insole
  Arms: 01
Device: Current standard of care insole — Current Medicare approved A5513 insole
  Arms: 02

SUMMARY:
To assess the efficacy of TrueContour® Insoles versus the current standard of care insoles in recurrence of plantar MTH ulcers in men and women, 18 years of age or older at the time of consent with clinical diagnosis of Diabetes Mellitus type 1 or type 2 who have had at least one recently healed plantar MTH foot ulcer (>1 week but <12 weeks since heeling) and have Loss of Protective Sensation.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, 18 years of age or older at the time of consent;
2. Clinical diagnosis of Diabetes Mellitus ;
3. At least one recently healed plantar MTH-related foot ulcer (>1 week but 4 months since heeling), based on medical records or if these cannot be obtained to the subject's best recollection OR current or recurring hemorrhage into callus under at least one MTH in a patient with a prior MTH related plantar ulcer that has been documented in the medical record;
4. Barefoot plantar pressure in the area of the previous MTH-related ulcer or at the area of current hemorrhagic callus >450 kPa;
5. Loss of Protective Sensation (refer to Section 7.2.6);
6. Community ambulator defined as having the ability or potential for ambulation outside in the community including the ability to traverse low-level environmental barriers such as curbs, stairs, or uneven surfaces, or better by subject report;
7. Ability to give consent;
8. In the opinion of the site PI the subject is willing and able to comply with the scheduled visits, treatment plan, and other trial procedures for the duration of the study.

Exclusion Criteria:

1. Presence of a current ulcer (see Section 7.1.1) below the malleoli, in the opinion of the site PI;
2. Partial foot amputation greater than of two metatarsal heads or rays per foot; toe amputations with the metatarsal heads left in place are permissible; complete foot amputation on one side (i.e. ambulation with a prosthesis) is permissible;
3. Charcot process that is active in the opinion of the site PI (requires immobilization beyond use of footwear that would be available through the study);
4. A prior ulcer on the plantar aspect of the heel within the last year, to the subject's best recollection that in the opinion of the site PI has high probability of recurring in the study footwear;
5. A prior ulcer on the weightbearing aspect of any toe within the last year, to the subject's best recollection that in the opinion of the site PI has high probability of recurring in the study footwear;
6. A prior ulcer on the plantar aspect of the foot associated with a mid-foot prominence at any time in the past, to the subject's best recollection that in the opinion of the site PI has high probability of recurring in the study footwear;
7. A prior ulcer on the plantar aspect of the foot associated with a mid-foot prominence at any time in the past, if the associated plantar pressure is >450kPa
8. Barefoot plantar pressure in the mid-foot that exceeds forefoot peak plantar pressure;
9. Need for an ankle-foot orthoses in the opinion of the site PI or another provider;
10. Need for more complex intervention, i.e. the site PI's decision is that the study footwear would not be adequate for the subject's needs, e.g. a rigid outsole or custom molded shoes are deemed necessary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The first occurrence of a plantar ulcer or pre-ulcer in subjects who have had one previously healed plantar ulcer | every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Loomis, MS, Principal Investigator — DIApedia, LLC
Locations (11):
- United States (11):
  - Carl T Hayden VA Medical Center, Phoenix, Arizona
  - Southern Arizona Limb Salvage Alliance, Tucson, Arizona
  - Center for Clinical Research, Inc, Castro Valley, California
  - Innovative Medical Technologies, Los Angeles, California
  - Diabetic Foot and Wound Center, Denver, Colorado
  - Weil Foot & Ankle Institute, Des Plaines, Illinois
  - Hines VA Hospital, Hines, Illinois
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Blair Medical Associates, Inc, Altoona, Pennsylvania
  - Temple University School of Podiatric Medicine, Philadelphia, Pennsylvania
  - Complete Family Footcare, McAllen, Texas

REFERENCES:
- [Derived] Ulbrecht JS, Hurley T, Mauger DT, Cavanagh PR. Prevention of recurrent foot ulcers with plantar pressure-based in-shoe orthoses: the CareFUL prevention multicenter randomized controlled trial. Diabetes Care. 2014 Jul;37(7):1982-9. doi: 10.2337/dc13-2956. Epub 2014 Apr 23. PMID 24760263